CLINICAL TRIAL: NCT06748209
Title: Portable Transcranial Magnetic Stimulation (TMS) in a Van for Treatment-Resistant Depression
Brief Title: Establishing Mobile Transcranial Magnetic Stimulation
Acronym: TMS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mark George, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00139739
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Major Depression
Keywords: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Mobile TMS qualifies as a Phase IV trial because it assesses the real-world efficacy of TMS therapy when administered via a mobile unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Open label Clinical TMS for Depression (Other): This will be FDA approved Left Prefrontal TMS for treating depression, we will be performing this within a VA, located at clinics throughout SC.
  Interventions: Device: Left prefrontal Transcranial Magnetic Stimulation (TMS); Device: FDA cleared TMS for treating depression

INTERVENTIONS:
Device: Left prefrontal Transcranial Magnetic Stimulation (TMS) — FDA cleared TMS
Device: FDA cleared TMS for treating depression — This is FDA approved TMS

SUMMARY:
In this pilot study, investigators propose to design and create a portable TMS unit, in a van, and then test out delivering TMS in three different locations in South Carolina, all affiliated with MUSC and within 2-hours driving from Charleston, SC. This study would test out this new delivery mode, and provide valuable feasibility, safety, and efficacy lessons for later refinement and potential widespread adoption of mobile TMS as a treatment option, both in our state and across the US.

DETAILED DESCRIPTION:
In this pilot study, investigators propose to design and create a portable TMS unit, in a van, and then test out delivering TMS in three different locations in South Carolina, all within 90 minutes driving from Charleston, SC. This study would test out this new delivery mode, and provide valuable lessons for later refinement and potential widespread adoption of mobile TMS as a treatment option. This would open up access to TMS for millions of patients with treatment resistant depression who cannot be treated in the current model. After this pilot feasibility and efficacy study, future research would use mobile TMS units for siting at residential care facilities, or remote hospitals and clinics.

Investigators aim to determine whether it is possible to assemble and build a functioning mobile TMS unit. After assembling the van, investigators will then recruit up to 30 treatment-resistant depression patients who live near one of three satellite MUSC clinics. These clinics are all within a 2 hour drive from the MUSC Charleston campus. Investigators will treat these patients, open label, with FDA approved accelerated TMS (6 sessions each day, over 2 hours, for 5 days, spread over one or two weeks). Investigators will measure TMS effectiveness using standard depression rating scales. Importantly, investigators will also collect the costs of performing the TMS which will inform whether MUSC or other health delivery systems might adopt this TMS method.

ELIGIBILITY:
Inclusion Criteria:

* Adult (22-80 years old)
* Have treatment-resistant depression as defined by the e-Mini, and the antidepressant treatment history form (ATHF short).
* Be able to read and communicate in English.
* Able to provide their own consent.
* Access to a computer with videoconferencing ability for initial consent and telescreen.

Exclusion Criteria:

* Patients with unstable medical conditions that might make TMS unsafe. This includes current poorly controlled seizures.
* Ferromagnetic metal in the head.
* Pregnant.
* Currently active substance abuse except tobacco.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of depression responders | From baseline to 1 week immediately after treatment week
  Number of patients with >50% improvement in Phq-9 scores before and then after 5 days of treatment
Improvement in Depression Symptoms | From baseline to 1 week immediately after treatment week
  Change in Phq-9 ratings from baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univerity of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
age, gender, degree of treatment resistance, current medications, changes in depression scores
Supporting Information: Study Protocol, ICF
Time Frame: After conclusion of the study and for 5 years after publication.
Access Criteria: All credible investigators, by writing and asking permission from the study PI and team.
URL: https://scresearch.org/studies/search?utf8=%E2%9C%93&q=Mark+George&commit=GO